CLINICAL TRIAL: NCT04908124
Title: An Open Label, Parallel-design, Clinical Investigation to Determine the Effectiveness and Safety of Five Water Based Personal Lubricants for the Relief of Intimate Discomfort Associated With Vaginal Dryness.
Brief Title: A Clinical Investigation Into the Effectiveness and Safety of Five Water Based Personal Lubricants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5025002
Record Dates: First submitted 2021-03-30; First posted 2021-06-01 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-02

CONDITIONS: Dyspareunia; Vaginal Dryness
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Intervention Model Description: The personal lubricants will be tested in a 5-arm parallel-design, where subjects will be randomised to an arm/lubricant. This follows an initial tolerance phase conducted in a sub-set of the population which will be tested in a 5-arm parrallel design,where subjects will be randomised to an arm/lubricant. Note: subjects participating in the both the tolerability and treatment phases will be enrolled into an arm for each which includes the same IP/lubricant throughout both phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Lubricant A - Tolerance (Experimental): A 3-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment.
  This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Interventions: Device: Lubricant A
- Lubricant B - Tolerance (Experimental): A 3-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment.
  This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Interventions: Device: Lubricant B
- Lubricant C - Tolerance (Experimental): A 3-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment.
  This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Interventions: Device: Lubricant C
- Lubricant D - Tolerance (Experimental): A 3-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment.
  This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Interventions: Device: Lubricant D
- Lubricant E - Tolerance (Experimental): A 3-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment.
  This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Interventions: Device: Lubricant E
- Lubricant A - Treatment (Experimental): A 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  This includes a sub-set population who were also enrolled into the arm using the same IP for the tolerability phase.
  Interventions: Device: Lubricant A
- Lubricant B - Treatment (Experimental): A 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  This includes a sub-set population who were also enrolled into the arm using the same IP for the tolerability phase.
  Interventions: Device: Lubricant B
- Lubricant C - Treatment (Experimental): A 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  This includes a sub-set population who were also enrolled into the arm using the same IP for the tolerability phase.
  Interventions: Device: Lubricant C
- Lubricant D - Treatment (Experimental): A 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  This includes a sub-set population who were also enrolled into the arm using the same IP for the tolerability phase.
  Interventions: Device: Lubricant D
- Lubricant E - Treatment (Experimental): A 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  This includes a sub-set population who were also enrolled into the arm using the same IP for the tolerability phase.
  Interventions: Device: Lubricant E

INTERVENTIONS:
Device: Lubricant A — Water-based lubricant, which is suitable for oral, anal and vaginal sexual intercourse. Approximately 3g of lubricant will be considered a single application.
  Other Names: Durex Play Feel
  Arms: Lubricant A - Tolerance; Lubricant A - Treatment
Device: Lubricant B — Water-based lubricant, which is suitable for oral, anal and vaginal sexual intercourse. Approximately 3g of lubricant will be considered a single application.
  Arms: Lubricant B - Tolerance; Lubricant B - Treatment
Device: Lubricant C — Water-based lubricant, which is suitable for oral, anal and vaginal sexual intercourse. Approximately 3g of lubricant will be considered a single application.
  Other Names: Durex Naturals Moisture
  Arms: Lubricant C - Tolerance; Lubricant C - Treatment
Device: Lubricant D — Water-based lubricant, which is suitable for oral, anal and vaginal sexual intercourse. Approximately 3g of lubricant will be considered a single application.
  Arms: Lubricant D - Tolerance; Lubricant D - Treatment
Device: Lubricant E — Water-based lubricant, which is suitable for oral, anal and vaginal sexual intercourse. Approximately 3g of lubricant will be considered a single application.
  Arms: Lubricant E - Tolerance; Lubricant E - Treatment

SUMMARY:
This clinical investigation will look at the safety of five water based personal lubricants, and teir effectiveness the relief of intimate discomfort associated with vaginal dryness.

DETAILED DESCRIPTION:
This is an open label, five-arm, parallel-design clinical investigation determining the effectiveness and safety of five personal lubricants. This clinical investigation consists of two phases, a Tolerance Phase and a Treatment Phase, whereby a sub-set of subjects will enter both the Tolerance Phase followed by the Treatment Phase. The remaining subjects will enter the Treatment Phase only.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is female and aged: 18 years to 65 years.
3. Female subject in a mutually monogamous heterosexual relationship (≥ 3 months) who is sexually active, defined as having sexual intercourse at least once a week.
4. Female subject of childbearing potential who is willing to use a highly effective method of contraception throughout the clinical investigation.
5. Female subject that agrees to have a gynaecological pelvic examination to ensure no significant disease findings and have intact skin and mucous in the test region assessed by the gynaecologist at all the relevant time points.
6. Subjects reporting mild to moderate vaginal dryness and dyspareunia during sex (when not using lubricant) in the past 3 months as confirmed on the Verbal Rating Scale (VRS).

Post-menopausal Inclusion Criteria:

1. Female subject in post-menopausal phase defined as having amenorrhea (absence of menstruation) for at least 12 months.
2. Female subject with premature menopause - surgical menopause or physiological menopause within the last 12 months or after having received chemotherapy.

Exclusion Criteria:

1. Female subject who is pregnant, breast-feeding or trying to conceive.
2. Female subject who has previously experienced an irritant or allergic reaction to any personal lubricant, vaginal moisturiser or female hygiene product or known to suffer from any contact allergen and/or are allergic to the investigational product ingredients.
3. Female subject has urinary, vaginal infection (fungal, bacterial) or sexually transmitted infection as diagnosed by the investigator.
4. Female subject presenting signs of internal irritation, active psoriasis, eczema or other active skin disorder or with a history of skin disorder
5. Female subject presenting clinically abnormal findings other than irritation during the physical examination that will affect study outcome.
6. Female subject who has started, stopped or changed hormonal treatments (including contraceptives) during the previous 3 months prior to screening.
7. Female subject who has used any kind of topical histamine and/or topical hormonal based product for local treatment of vaginal dryness in the past 3 months.
8. Female subject with any medical conditions which in the opinion of the investigator could compromise the immune function.
9. Female subject taking steroid preparations, immune-suppressive drugs or any other medication which in the opinion of the investigator may affect the test results.
10. Female subject who has had any change to medication or treatment regimen for the treatment of diabetes mellitus during the previous 3 months prior to screening.
11. Female subject that will be unable to comply fully with the study requirements or unable to tolerate the procedures.
12. Female subject that have had a suspicion of malignancy or history of malignancy within the past 2 years.
13. Female subject who has had surgical cervical excision or vaginal and/or vulvar procedures in the previous year.
14. Female subject that has had a positive cervical screening examination for Human Papillomavirus (HPV) within the 3 years of the screening visit.
15. Female subject currently being treated with systemic medications or medicines that act locally in the vaginal area.
16. Female subject using vaginal douches and is unwilling to stop its use at least 2 weeks prior to screening and throughout the clinical investigation.
17. Female subject has changed contraceptive medication within the past 3 months or intending to change contraceptive medications.
18. Female subject has participated in another investigation within 3 months prior to screening.
19. Subject who is an employee at the site or a partner or first-degree relative of the Investigator.
20. Subject fails to satisfy the investigator of fitness to participate for any other reason.

Post-Menopausal Exclusion Criteria:

1. Female subject that has had previous episodes of vaginal bleeding of unknown origin within the last 6 months of the screening visit.
2. Female subject showing vaginal prolapse and/or other medical conditions that could interfere with the study conduct and participation.
3. Female subject that have used any kind of systemic and/or local hormonal products for the treatment of vaginal dryness or any other vaginal condition in the 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) score compared to baseline | 4 weeks after baseline
  The Change in FSFI from the baseline event and at 4-weeks post baseline

SECONDARY OUTCOMES:
Change from baseline in the Female Sexual Function Index (FSFI) individual domain scores | 4 weeks after baseline
  Change from baseline in the FSFI individual domain scores (desire, arousal, lubrication, orgasm, satisfaction, and pain) at 4-weeks post baseline
Overall proportion of subjects with Adverse Events/Adverse Device Effects (AE/ADEs) | 4 weeks
  Overall proportion of subjects with Adverse Events/Adverse Device Effects (AE/ADEs) i.e. the occurrence of one of more AE/ADE per subject.
Subject perception of the personal lubricants through Subject Percieved Questions | Initial application (within 24 hours of intercourse) and after 4 weeks
  Subjects' perception of each of the five personal lubricants will be determined through Subject Perceived Questions
Global evaluation of the personal lubricants (subjective opinion) | 4 weeks after baseline
  • Subjects global evaluation of the five personal lubricants will be determined through global evaluation of effectiveness, tolerability and usability
Vaginal Epithelial Tolerability (VET) | Baseline, 2 and 24 hours post single application
  An assessment of the Vaginal Epithelial Tolerability (VET) of the five personal lubricants as assessed by gynaecologist examination.
Tolerability as assessed by Subject Perceived Questions | 24 hours post single application.
  Tolerability of the five personal lubricants will be determined through Subject Perceived Questions
Global Assessment of Tolerance for each subject by a Gynaecologist | 24 hours post single application
  Determined by professional assessment of each individual.
Overall Tolerance Rating Statement for each lubricant by a Gynaecologist | 24 hours post single application
  An overall summary statement of tolerance of each lubricant will be made by the Gynaecologist, taking into consideration all tolerance assessments across all subjects and the nature of the IP in its intended use

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Dr., Principal Investigator — proDERM GmbH
Locations (1):
- proDERM GmbH, Hamburg, Pinneberg, Germany

IPD SHARING:
Plan to Share IPD: No